CLINICAL TRIAL: NCT04814524
Title: A Digital Intervention Protocol to Enhance Recovery After Head and Neck Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ryan Li, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00021902; NCI-2020-11592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00021902 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Head and Neck Carcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (VR, Fitbit) (Experimental): Beginning postoperative day 1, patients use VR over 30 minutes up to 4 times daily on weekdays and 2 times daily on weekends, and wear Fitbit daily with a goal of 2,000 steps until the day of discharge, or until 14 days after surgery. Pre and post-VR pain scores will be obtained for each VR use. Sleep data may also be evaluated from Fitbit devices.
  Interventions: Device: Fitbit; Other: Questionnaire Administration; Device: Virtual Reality Device
- Group 2 (VR) (Experimental): Beginning postoperative day 1, patients use VR over 30 minutes up to 4 times daily on weekdays and 2 times daily on weekends until the day of discharge or until 14 days after surgery. Pre and post-VR pain scores will be obtained for each VR use.
  Interventions: Other: Questionnaire Administration; Device: Virtual Reality Device
- Group 3 (Fitbit) (Experimental): Beginning postoperative day 1, patients wear Fitbit daily with a goal of 2,000 steps until the day of discharge or until 14 days after surgery. Sleep data may also be evaluated from Fitbit devices.
  Interventions: Device: Fitbit; Other: Questionnaire Administration
- Group 4 (questionnaire) (Active Comparator): Patients do not use VR or wear Fitbit.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Device: Fitbit — Wear Fitbit
  Arms: Group 1 (VR, Fitbit); Group 3 (Fitbit)
Other: Questionnaire Administration — Ancillary studies
Device: Virtual Reality Device — Use VR
  Arms: Group 1 (VR, Fitbit); Group 2 (VR)

SUMMARY:
This trial studies examines the impact of virtual reality (VR) experiences and Fitbit wearable activity devices on postoperative recovery after head and neck surgery. Virtual reality has shown to help rehabilitation and pain control primarily in non-surgical fields, and researchers are interested in using this to help postoperative pain control. Early mobilization after surgery is also important, and may increase lung capacity, improve gastrointestinal function, reduce pain, and reduce risk of deep venous thrombosis. Use of virtual reality and Fitbit devices may improve postoperative pain control and reduce narcotic use among hospitalized patients after head and neck surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the effectiveness of daily virtual reality (VR) therapy during hospitalization, compared to patients not utilizing daily VR therapy.

II. Evaluate the effectiveness of daily ambulation goals using Fitbit devices during hospitalization, compared to patients without daily ambulation goals.

III. Evaluate the effectiveness of daily VR use and daily Fitbit ambulation goals during hospitalization.

EXPLORATORY OBJECTIVES:

I. Evaluate the effectiveness of daily VR use and daily Fitbit ambulation goals during hospitalization on reducing pain scores, anxiety, depression, and length of stay, and improving sleep quality, hospital satisfaction, and disposition on discharge.

OUTLINE: Patients are randomized to 1 of 4 groups.

GROUP 1: Beginning postoperative day 1, patients use VR over 30 minutes up to 4 times daily on weekdays and 2 times daily on weekends, and wear Fitbit daily with a goal of 2,000 steps until the day of discharge, or until 14 days after surgery. Pre and post-VR pain scores will be obtained for each VR use. Sleep data may also be evaluated from Fitbit devices.

GROUP 2: Beginning postoperative day 1, patients use VR over 30 minutes up to 4 times daily on weekdays and 2 times daily on weekends until the day of discharge or until 14 days after surgery. Pre and post-VR pain scores will be obtained for each VR use.

GROUP 3: Beginning postoperative day 1, patients wear Fitbit daily with a goal of 2,000 steps until the day of discharge or until 14 days after surgery. Sleep data may also be evaluated from Fitbit devices.

GROUP 4: Patients do not use VR or wear Fitbit.

ELIGIBILITY:
Inclusion Criteria:

* English speaking (Ability to interact with virtual reality content may be impacted by inability to understand English)
* Older than 18 years of age and younger than 89 years of age. Both men and women and members of all races and ethnic groups will be included
* Planned to undergo major surgery at Oregon Health & Science University (OHSU) with the Department of Otolaryngology-Head and Neck Surgery with an expected length of stay (LOS) of 2 days or more
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Planned postoperative admission to the intensive care unit (ICU)
* Social or psychiatric conditions that may interfere with compliance
* Isolation precautions
* Complex head and neck procedure requiring resection or reconstruction involving the scalp, orbit, or mid-face. This would limit the ability to utilize the VR headset
* Reconstruction, incisions, wounds, wound care, or injury that impact the ability to place on the VR headset or wear a Fitbit device around the wrist. This would limit the ability to utilize the VR headset or the Fitbit device
* History of seizure or epilepsy
* History of vertigo or persistent dizziness
* Use of cardiac pacemaker, requirement for hearing aid on at all times, or have defibrillators
* Limitations that impair mobility. This would limit the ability to utilize the Fitbit device
* Use of a walker or wheelchair at baseline. This would limit the ability to utilize the Fitbit device
* Children
* Pregnant women
* Neonates of uncertain viability or nonviable neonates
* Decisionally impaired adults
* Prisoners

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Mean daily opioid use | Through study completion, an average of 10 days
  Will be assessed using milligram morphine equivalents (MME). Narcotic use may be compared using One-Way Analysis of Variance (ANOVA) and two sample t-test can be used to compare the narcotic use between intervention group and control group (virtual reality [VR]+Fitbit versus [vs.] control, VR vs. control, Fitbit vs. control). Furthermore, a linear regression model including demographic and clinical characteristic variables with a P-value =< 0.1 will be used to determine factors associated with reduced narcotic use.

OTHER OUTCOMES:
Pain scores | Through study completion (pre and post-VR use), an average of 10 days
  Will review the electronic medical record (EMR) to evaluate daily pain scores among patients, and average these scores to obtain the daily pain score. May also look at differences between AM and PM pain scores among the different cohorts. Additionally, we plan to evaluate pain scores obtained pre and post-VR use. Descriptive statistics can be used to present the results of anxiety. One-way ANOVA and two-sample t-test can be used to compare differences between the groups.
Anxiety | Before surgery and at study completion, an average of 10 days
  Will use the Generalized Anxiety Disorder 7-Item scale to determine preoperative and postoperative level of anxiety. Scores may represent mild (6-10), moderate (11-15), and severe (16-21) anxiety. Descriptive statistics can be used to present the results of anxiety. One-way ANOVA and two-sample t-test can be used to compare differences between the groups.
Depression | Before surgery and at study completion, an average of 10 days
  Will use the Patient Health Questionaire-9 to determine preoperative and postoperative level of depression. This is a screening instrument with 9 items that measures depression, with answers as not at all, several days, more than half of the days, and nearly every day (score 0-27). Scores may represent mild (5-9), moderate (10-19), and severe (>= 20) depression. Descriptive statistics can be used to present the results of depression. One-way ANOVA and two-sample t-test can be used to compare differences between the groups.
Sleep quality | Before surgery and at study completion, an average of 10 days
  Will use the Insomnia Severity Index to determine preoperative and postoperative sleep quality. Items are rated on a 5-point Likert scale, and a total score ranges from 0 to 28. Scores may represent subthreshold (8-14), moderate (15-21), or severe (22-28) insomnia. Descriptive statistics can be used to present the results of sleep quality. One-way ANOVA and two-sample t-test can be used to compare differences between the groups.
Sleep patterns | At study completion, an average of 10 days
  Will evaluate sleep patterns among patients with Fitbit devices to better understand inpatient sleep in the hospital. Descriptive statistics can be used to present the results of LOS. One-way and two-sample t-test can be used to analyze differences between the groups.
Hospital satisfaction | At study completion, an average of 10 days
  Will use a Visual Analogue Scale to analyze patient satisfaction during hospitalization, and which would be provided to patients on day of discharge. The Visual Analogue Scale (VAS) is a horizontal line that is 100-mm long, with no satisfaction (0) on the very left and extreme satisfaction on the very right (100). Descriptive statistics can be used to present the results of hospital satisfaction. One-way ANOVA and two-sample t-test can be used to compare differences between the groups.
Disposition on discharge | At study completion, an average of 10 days
  Will evaluate data regarding disposition on discharge to home, home with home health, skilled nursing facility, inpatient rehabilitation facility, remain in hospital, other facility, or remaining in the hospital from the EMR on the day of discharge or day 14 of hospital stay. Descriptive statistics can be used to present the results of disposition on discharge. Chi-square test can be used to compare differences between the groups.
Length of stay (LOS) | At study completion, an average of 10 days
  Will determine LOS beginning from postoperative day one and to include the day of discharge. Descriptive statistics can be used to present the results of LOS. One-way ANOVA and two-sample t-test can be used to analyze differences between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Li, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States